CLINICAL TRIAL: NCT06309173
Title: Development of Digital Biomarkers in Multiple Sclerosis: Validation Study 2
Acronym: DreaMS_VS2
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 0000-00000; ko23Hemkens
Record Dates: First submitted 2024-03-06; First posted 2024-03-13 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-09

CONDITIONS: Multiple Sclerosis
Keywords: Digital Biomarkers
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Multiple sclerosis (MS) is a chronic inflammatory disease of the central nervous system (CNS). Diagnosis is established by clinical assessment of persons with MS (PwMS), in combination with imaging and body fluid assessments. Treatment decisions in MS are mainly based on periodic monitoring of disease activity and progression through clinical and imaging assessments.

The predictive and prognostic value of currently used assessments to individualize treatment decisions is still very limited. Emerging digital measures have the potential to provide granular health status measurements that would allow monitoring MS disease activity and progression continuously and remotely, in real-world settings, with minimal disruption of patients' life.

Using the investigators' self developed dreaMS software program the investigators previously identified digital biomarkers (DB) that hold promise to provide detailed and accurate assessments of MS-related health status and disease progression to complement traditional clinical, imaging, or body fluid assessments.

This international, observational study aims to evaluate and validate the generalizability of these DB across different languages and cultural settings to provide DB that are helpful for patient care, research, and regulatory decisions. Beyond this, the processes and data structures created for this study are intended to establish a collaborative research platform for subsequent studies, including pragmatic trials, promoting new long-term international academic collaborations.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is a chronic inflammatory disease of the central nervous system. Focal demyelination and diffuse neurodegeneration in the gray and white matter of the brain and spinal cord lead to decreased physical and cognitive functioning and disability.

Diagnosis is established by clinical assessment of persons with MS (PwMS), including taking their history and neurologic examination, in combination with imaging and body fluid assessments. Treatment decisions in MS are based on continuous monitoring of MS disease activity and progression through clinical and imaging assessments, while the role of body fluid assessments is not yet universally established. The predictive and prognostic value of these currently used assessments to individualize treatment decisions is still very limited. New and more reliable measures are needed, especially indicators of disease progression, which allow to personalize therapies and care.

With the digitization of healthcare, new opportunities are emerging to provide quasi-continuous and granular health status measurements as digital measures. Such digital measures may allow to monitor MS disease activity and progression more informatively than the only episodical traditional assessments. Digital health technologies allow to remotely capture dynamic fluctuating functions and symptoms in real world settings with minimal disruption of patients' life and usual care.

The investigators developed the dreaMS software program that includes app-based interactions with the patients, patient-reported information via surveys, and continuous monitoring through sensors. In a previous study (NCT04413032), which evaluated the feasibility and acceptance of using our dreaMS software program, we identified digital biomarkers (DB) that are relevant for PwMS. These DB are evaluated and validated in an ongoing study including a larger population of PwMS in Switzerland (NCT05009160).

This international, observational study aims to evaluate and validate the generalizability of these DB across different languages and cultural settings to provide DB that are helpful for patient care, research, and regulatory decisions. Beyond this, the processes and data structures created for this study are intended to establish a collaborative research platform for subsequent studies, including pragmatic trials, promoting new long-term international academic collaborations.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18
* Diagnosed with MS according to the revised McDonald criteria 2017, all clinical forms inclusive (CIS, RRMS, SPMS, PPMS)
* In possession of a Healios+Me app-compatible smartphone (iOS/Android)
* Corrected close visual acuity of ≥0.5
* Hand motor skills sufficient for using a smartphone
* Ability and intention to follow the study procedures
* Sufficient knowledge of the language for the specific country
* Informed Consent as documented by signature

Exclusion Criteria:

* NA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Persons with MS from the neurological outpatient clinics in the participating centers (European and North American).
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Correlation of the digital features with the respective measurements of the clinical reference tests | Baseline, 12 months, 24 months
  Spearman correlation coefficients higher than 0.4 (lower bound of 95% confidence interval) are considered relevant. All scheduled pairs of measurements collected during the study will be used. As the yearly observations of a patient are not independent, standard conﬁdence intervals cannot be used. Therefore, a bootstrap approach will be used to determine a 95% conﬁdence interval for the Spearman correlations (where data will be resampled on the patient level).
The ability of measurements of the changes in the digital biomarkers over the two-year follow-up to predict worsening in the clinical reference test over the same period expressed as binary variables | Baseline and 24 months
  The change of the digital biomarker over two years allows to distinguish patients experiencing a relevant worsening in the corresponding reference test over the same period from those who do not with an area under the receiver operating characteristic curve (AUC) larger than 0.6 (lower bound of 95% confidence interval).

SECONDARY OUTCOMES:
The ability of the digital biomarker to detect worsening in other relevant reference test results creating converging evidence | up to 24 months
  The ability of the digital biomarker to detect worsening in other relevant reference test results creating converging evidence
The ability of the digital biomarker to detect worsening in standard assessments used for treatment of PwMS (clinical, imaging, body fluids) | up to 24 months
  The ability of the digital biomarker to detect worsening in standard assessments used for treatment of PwMS (clinical, imaging, body fluids)
The ability of the digital biomarker to detect change of Patient Reported Outcomes | up to 24 months
  The ability of the digital biomarker to detect change of Patient Reported Outcomes
The ability of the digital biomarker to detect occurrence of clinical and other meaningful events (relapses, PIRA, serious adverse events, hospitalizations, working capacity) | up to 24 months
  The ability of the digital biomarker to detect occurrence of clinical and other meaningful events (relapses, PIRA, serious adverse events, hospitalizations, working capacity)
The relationship of the digital biomarkers with imaging and body fluid markers | up to 24 months
  The relationship of the digital biomarkers with imaging and body fluid markers
The relationship of the digital biomarkers with Patient Reported Outcomes | up to 24 months
  The relationship of the digital biomarkers with Patient Reported Outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Ludwig Kappos, Prof., Study Director — University Hospital, Basel, Switzerland
Locations (3):
- University of California, San Francisco (UCSF) Weill Institute, Department of Neurology, San Francisco, California, United States
- Austria (2):
  - Innsbruck Medical University, Department of Neurology, Innsbruck, Tyrol
  - Vienna Medical University, Department of Neurology, Vienna

IPD SHARING:
Plan to Share IPD: Undecided